CLINICAL TRIAL: NCT04475601
Title: A Prospective, Multicenter, Randomized PHASE II Clinical Trial of Enzalutamide Treatment to Decrease the Morbidity in Patients With Corona Virus Disease 2019 (COVID-19)
Brief Title: Enzalutamide Treatment in COVID-19
Acronym: COVIDENZA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: By sponsor, based on DSMB recommendations
Sponsor: Andreas Josefsson (Other Government)
Collaborators: Umeå University (Other); Sahlgrenska University Hospital (Other); University Hospital, Umeå (Other); Uppsala University Hospital (Other); Skane University Hospital (Other); Jonkoping County Hospital (Other); Sundsvall Hospital (Other); Helsingborgs Hospital (Other); Göteborg University (Other); Astellas Pharma Europe Ltd. (Industry); Norrlands University Hospital (Other)
Responsible Party: Sponsor-Investigator, Andreas Josefsson, Assistant Professor and Consultant Urologist, Region Västerbotten
Organization: Region Västerbotten (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVIDENZA
Record Dates: First submitted 2020-06-08; First posted 2020-07-17 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2021-08

CONDITIONS: COVID-19; Corona Virus Infection
Keywords: Enzalutamide; Randomized clinical trial; COVID-19; Sars-CoV2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — enzalutamide

STUDY DESIGN:
Intervention Model Description: Prospective, randomized (2:1), open, multicentre, clinical controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enzalutamide+Standard of Care (Experimental): Up to 5 days with 4x40 mg enzalutamide tablets orally once daily
  Interventions: Drug: Enzalutamide Pill
- Standard of Care (No Intervention): Standard of care

INTERVENTIONS:
Drug: Enzalutamide Pill — The once daily dose will be given only during hospitalization and stop if starting invasive mechanical ventilation or at discharge from hospital
  Arms: Enzalutamide+Standard of Care

SUMMARY:
COVID-19 is a disease with high rate of morbidity if symptomatic. There is a great need of treatments to decrease the severity. The vast majority of patients needing intensive care are men, and this may be due to the androgens, either by regulation of TMPRSS2, necessary for virus internalization, or other mechanisms. Enzalutamide is an antiandrogen inhibiting the expression of androgen regulated proteins, such as TMPRSS2. The aim of this trial is to evaluate a possible beneficial effect of short-term enzalutamide treatment of COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID-19 test
* Mild to severe symptoms of COVID-19
* Hospitalization
* WHO performance status 0-3
* Age above or equal to 50 years
* Can understand all the requirements of the study, provide informed consent, and provide authorization of use and disclosure of personal health information.
* Estimated expected survival of 1 year (excluding symptoms due to COVID-19)

Exclusion Criteria:

* Severe allergy to Enzalutamide
* Pregnant or breast-feeding women
* Need of immediate mechanical ventilation
* Current medication includes enzalutamide treatment
* Stroke or Transitory Ischemic attack in medical history
* Treatment for HIV
* Treatment with tamoxifen
* Treatment with immunosuppressive agents
* Severe immunosuppressive disease
* Treatment with warfarin or NOAC (Non-vitamin K-antagonist anticoagulants)
* Previous seizure in medical history
* Other serious illness or medical condition
* Unstable cardiovascular disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Time to worsening of disease | Up to 30 days after inclusion
  Clinical worsening to invasive mechanical ventilation or death as assessed by the 7-point ordinal scale
Time to improvement of disease | Up to 30 days after inclusion
  Time to discharge from hospital assessed by the 7-point ordinal scale

SECONDARY OUTCOMES:
Adverse events | Up to 6 months
  Safety evaluation, as measured by AEs
Duration of supplemental oxygen (days) | Up to 30 days
  Total days of extra oxygen
Admission to ICU | Up to 30 days and up to 6 months
  Frequence of admission to ICU
Laboratory assessment of Hemoglobin concentration day 0, 2, 4 and 6 | Up to 30 days
  Changes of laboratory parameters: Hb
Virus load assessment day 0, 2, 4 and 6 | UP to 7 days
  PCR based SARS-CoV-2 measurement from upper respiratory tract
Hospital stay (days) | Up to30 days and 6 months
  Total number of days evaluated at 30 days and 6 months
Re-admission to hospital due to rebound COVID-19 | Evaluated for 30 days and after 6 months
  If admitted to hospital due to COVID-19 disease after discharge from hospital
Mortality at 6 months | up to 30 days and up to 6 months respectively
  Death due to any cause
Laboratory assessment of CRP concentration day 0, 2, 4 and 6 | Up to 30 days
  Changes of laboratory parameters: CRP
Laboratory assessment of liver function day 0, 2, 4 and 6 | Up to 30 days
  Changes of laboratory parameters: ALAT, ASTA and/or ALP
Laboratory assessment of creatinine concentration day 0, 2, 4 and 6 | Up to 30 days
  Changes of laboratory parameters: Createnin
Laboratory assessment of D-dimer concentration day 0, 2, 4 and 6 | Up to 30 days
  Changes of laboratory parameters: D-dimer
Laboratory assessment of platelets concentration day 0, 2, 4 and 6 | Up to 30 days
  Changes of laboratory parameters: TPK
Laboratory assessment of IL-6 concentration day 0, 2, 4 and 6 | Up to 30 days
  Changes of laboratory parameters: IL-6
Laboratory assessment of B- and T-lyphocytes concentration day 0, 2, 4 and 6 | Up to 30 days
  Changes of laboratory parameters: Differentiate count of leucocytes
Pharmacokinetic interaction of enzalutamide with steroids | Up to 30 days
  Maximum Plasma Concentration [Cmax] of steroids in blood

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Josefsson, MdPhD, Principal Investigator — Norrlands University Hospital, Region Västerbotten
Locations (6):
- Sweden (6):
  - Anders Bjartell, Malmo, Skåne County
  - Ryhovs Hospital, Jönköping, Småland
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Sundsvall Region Hosptial, Sundsvall
  - Umeå Univerisity Hospital, Umeå

IPD SHARING:
Plan to Share IPD: Undecided
The extent of sharing will be regulated during the trial to consider the integrity of the data according GDPR and national laws

REFERENCES:
- [Derived] Welen K, Overby AK, Ahlm C, Freyhult E, Robinsson D, Henningsson AJ, Stranne J, Bremell D, Angelin M, Lindquist E, Buckland R, Carlsson CT, Pauksens K, Bill-Axelsson A, Akre O, Ryden C, Wagenius M, Bjartell A, Nilsson AC, Styrke J, Repo J, Balkhed AO, Niward K, Gisslen M, Josefsson A. COVIDENZA - A prospective, multicenter, randomized PHASE II clinical trial of enzalutamide treatment to decrease the morbidity in patients with Corona virus disease 2019 (COVID-19): a structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Mar 16;22(1):209. doi: 10.1186/s13063-021-05137-4. PMID 33726804
- See also: Publication of the results — https://doi.org/10.1016/j.eururo.2021.12.013